CLINICAL TRIAL: NCT01271985
Title: Fixed-dose Combination Therapy (PolyPill) in Primary and Secondary Prevention of Cardiovascular Disease in Middle-aged and Elderly Iranians
Brief Title: Prevention of Cardiovascular Disease in Middle-aged and Elderly Iranians Using a Single PolyPill
Acronym: PolyIran
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Golestan University of Medical sciences (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DDRC.89.17
Record Dates: First submitted 2010-12-14; First posted 2011-01-07 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Drug Combinations; prevention and control; Aspirin; Antihypertensive Agents; Antilipemic Agents
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Self-Care Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PolyPill (Active Comparator): PolyPill once daily and Minimal Care
  Interventions: Drug: PolyPill; Other: Minimal care
- Minimal care (Active Comparator): Minimal care.
  Interventions: Other: Minimal care
- Usual care (No Intervention): Basic primary health care provided by the local physicians and Community Health Workers consistent with the current Iranian Health Care System guidelines.

INTERVENTIONS:
Drug: PolyPill — A combination tablet containing Aspirin 81 mg, enalapril 5 mg (or valsartan 40 mg), atorvastatin 20 mg and hydrochlorothiazide 12.5 mg taken once daily
  Other Names: PolyPill 4-1; PolyPill 4-2
  Arms: PolyPill
Other: Minimal care — Health education pamphlet on reducing cardiovascular risk factors, direct education on reducing cardiovascular risk factors provided by the study physician and the Community Health Worker, biannual follow-up and BP measurement
  Arms: Minimal care; PolyPill

SUMMARY:
The purpose of this study is to determine the effects of PolyPill tablet (a fixed dose combination of two anti-hypertensive medications, atorvastatin and aspirin) on primary and secondary prevention of cardiovascular disease in Iranian adults older than 50.

DETAILED DESCRIPTION:
Cardiovascular diseases (myocardial infarction and stroke) are the most common cause of death and disability in Iran and account for nearly half of all-cause mortality in Iranians. Therefore, prevention of cardiovascular diseases is a top priority in countries with limited health system budgets such as Iran.

Eighty seven to hundred percent of patients dying from Coronary Heart Disease (CHD) have at least one risk factor for cardiovascular diseases. Therefore, risk factor modification in middle-aged and old individuals might prevent death and is a main priority. Combination drug therapy has been proposed as a cost-effective measure to reduce modifiable risk factors for cardiovascular disease in aged people. It has been showed that combination drug therapy can potentially decrease ischemic heart events and strokes by 88 and 80 percent, respectively.

The purpose of this study is to determine the effects of PolyPill tablet (a fixed dose combination of two anti-hypertensive medications, atorvastatin and aspirin) on primary and secondary prevention of cardiovascular disease in Iranian adults older than 50.

This is a study on subjects older than 50 enrolled in the Golestan Cohort Study. The study is designed as a pragmatic cluster randomized trial. The study comprises three arms as follows:

1. 4234 randomly selected participants receive PolyPill tablets once daily and Minimal care (which consists of direct education and pamphlet on cardiovascular risk reduction, biannual follow-ups and BP measurements).
2. 4177 randomly selected participants receive only Minimal care as described above.
3. Include remaining 24000 participants of rural participants of Golestan cohort, aged 50 and higher who receive the basic primary health care provided by the local physicians and Community Health Workers for the whole participants of Golestan Cohort study consistent with the current Iranian Health Care System guidelines. A random sample of 4395 subjects from this usual care arm were selected from this group as the third arm of the study and outcome ascertainment will be performed for this sample and will be used in the secondary comparison.

Arms #1 and #2 are compared via a 2-armed open-labeled cluster Randomized Controlled Trial. Comparisons between arm #3 and the other 2 arms are also performed.

Endpoints include major cardiovascular events (death and hospitalization)

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years old
* Enrollment in the Golestan Cohort Study

Exclusion Criteria:

1. Hypersensitivity to any of PolyPill components:

   1. Hypersensitivity to Non-steroidal anti-inflammatory agents
   2. Hypersensitivity to statins
   3. Hypersensitivity to hydrochlorothiazide or sulfonamides
   4. Hypersensitivity to enalapril and valsartan
2. Past medical history of angioedema
3. Medical history of GI bleeding or peptic ulcer in the last 3 months
4. Pregnancy or lactation
5. Bleeding disorders such as hemophilia
6. Receiving anticoagulation therapy
7. Alcohol consumption greater than 40gr/week
8. Advanced liver disease
9. Uncontrolled seizures
10. Asthma with any of the following criteria present:

    1. Daily symptoms
    2. Asthmatic attacks waking the patient from sleep more than once a week
    3. History of nasal polyps
    4. Aspirin sensitive asthma
    5. Presence of rhinitis symptoms not due to infection
11. Past medical history of gout
12. Serum creatinine values above 2 mg/dL or a Glomerular Filtration Rate (GFR) below 30 mL/min
13. Hemoglobin concentrations below 11 g/dL for males and 10 g/dL for females
14. BP < 90/60
15. Debilitating medical/mental disorders affecting medication compliance (including psychosis, disabilities, and blindness)
16. Past medical history of stroke

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8410 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Time to first major cardiovascular event | 5 years
  Major cardiovascular events are defined as:
  1. Major coronary events include: sudden cardiac death, myocardial infarction, a diagnosis of angina, revascularization procedure
  2. Cerebrovascular accidents (CVA) including transient ischemic attacks (TIA)
  3. Hospitalization because of cardiovascular disease

SECONDARY OUTCOMES:
Blood pressure | 5 years
  Changes in blood pressure after 5 years
Fasting blood sugar, total cholesterol, HDL-C and LDL-C | 5 years
  Changes in fasting blood sugar and lipid profile after 5 years
Number of Subjects Developing Adverse Events | 5 years
  Number of participants who experience adverse effects to the PolyPill tablet leading to discontinuation.
Compliance | 5 years
  Compliance is measured by pill-count in participants of the intervention arm as percent pills taken.
Rate of major cardiovascular events | 5 years
  Number of major cardiovascular events (as described above) during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D., Study Chair — Digestive Disease Research Center
Locations (1):
- Golestan Cohort Study Center, Gonbad, Golestan Province, Iran

REFERENCES:
- [Background] Malekzadeh F, Marshall T, Pourshams A, Gharravi M, Aslani A, Nateghi A, Rastegarpanah M, Khoshnia M, Semnani S, Salahi R, Thomas GN, Larijani B, Cheng KK, Malekzadeh R. A pilot double-blind randomised placebo-controlled trial of the effects of fixed-dose combination therapy ('polypill') on cardiovascular risk factors. Int J Clin Pract. 2010 Aug;64(9):1220-7. doi: 10.1111/j.1742-1241.2010.02412.x. PMID 20653798
- [Background] Lonn E, Bosch J, Teo KK, Pais P, Xavier D, Yusuf S. The polypill in the prevention of cardiovascular diseases: key concepts, current status, challenges, and future directions. Circulation. 2010 Nov 16;122(20):2078-88. doi: 10.1161/CIRCULATIONAHA.109.873232. No abstract available. PMID 21098469
- [Background] Lonn E, Yusuf S. Polypill: the evidence and the promise. Curr Opin Lipidol. 2009 Dec;20(6):453-9. doi: 10.1097/MOL.0b013e32833305a3. PMID 19884824
- [Background] Malekzadeh F, Pourshams A, Marshall T. The preventive polypill--much promise, insufficient evidence. Arch Iran Med. 2007 Jul;10(3):430-1. No abstract available. PMID 17604490
- [Background] Majed M, Moradmand Badie S. A pilot double-blind randomised placebo-controlled trial of the effects of fixed-dose combination therapy ('polypill') on cardiovascular risk factors. Arch Iran Med. 2011 Jan;14(1):78-80. No abstract available. PMID 21194270
- [Background] PILL Collaborative Group; Rodgers A, Patel A, Berwanger O, Bots M, Grimm R, Grobbee DE, Jackson R, Neal B, Neaton J, Poulter N, Rafter N, Raju PK, Reddy S, Thom S, Vander Hoorn S, Webster R. An international randomised placebo-controlled trial of a four-component combination pill ("polypill") in people with raised cardiovascular risk. PLoS One. 2011;6(5):e19857. doi: 10.1371/journal.pone.0019857. Epub 2011 May 25. PMID 21647425
- [Background] Indian Polycap Study (TIPS); Yusuf S, Pais P, Afzal R, Xavier D, Teo K, Eikelboom J, Sigamani A, Mohan V, Gupta R, Thomas N. Effects of a polypill (Polycap) on risk factors in middle-aged individuals without cardiovascular disease (TIPS): a phase II, double-blind, randomised trial. Lancet. 2009 Apr 18;373(9672):1341-51. doi: 10.1016/S0140-6736(09)60611-5. Epub 2009 Mar 30. PMID 19339045
- [Background] Wald NJ, Law MR. A strategy to reduce cardiovascular disease by more than 80%. BMJ. 2003 Jun 28;326(7404):1419. doi: 10.1136/bmj.326.7404.1419. PMID 12829553
- [Background] Wald DS, Wald NJ. Implementation of a simple age-based strategy in the prevention of cardiovascular disease: the Polypill approach. J Eval Clin Pract. 2012 Jun;18(3):612-5. doi: 10.1111/j.1365-2753.2011.01637.x. Epub 2011 Jan 30. PMID 21276141
- [Background] Wald DS, Wald NJ. The Polypill in the prevention of cardiovascular disease. Prev Med. 2011 Jan;52(1):16-7. doi: 10.1016/j.ypmed.2010.11.015. Epub 2010 Dec 2. No abstract available. PMID 21130112
- [Background] Rifai L, Khan BV. Do the current medical and economic times dictate the need for the "polypill"? J Clin Hypertens (Greenwich). 2009 Dec;11(12):775-6. doi: 10.1111/j.1751-7176.2009.00188.x. No abstract available. PMID 20021541
- [Background] Soliman EZ, Mendis S, Dissanayake WP, Somasundaram NP, Gunaratne PS, Jayasingne IK, Furberg CD. A Polypill for primary prevention of cardiovascular disease: a feasibility study of the World Health Organization. Trials. 2011 Jan 5;12:3. doi: 10.1186/1745-6215-12-3. PMID 21205325
- [Background] Sepanlou SG, Poustchi H, Kamangar F, Malekzadeh R. Effectiveness and feasibility of lifestyle and low-cost pharmacologic interventions in the prevention of chronic diseases: a review. Arch Iran Med. 2011 Jan;14(1):46-53. PMID 21194261
- [Background] Sepanlou SG, Kamangar F, Poustchi H, Malekzadeh R. Reducing the burden of chronic diseases: a neglected agenda in Iranian health care system, requiring a plan for action. Arch Iran Med. 2010 Jul;13(4):340-50. PMID 20597569
- [Background] Sanz G, Fuster V. Fixed-dose combination therapy and secondary cardiovascular prevention: rationale, selection of drugs and target population. Nat Clin Pract Cardiovasc Med. 2009 Feb;6(2):101-10. doi: 10.1038/ncpcardio1419. Epub 2008 Dec 23. PMID 19104519
- [Background] Robinson JG, Maheshwari N. A "poly-portfolio" for secondary prevention: a strategy to reduce subsequent events by up to 97% over five years. Am J Cardiol. 2005 Feb 1;95(3):373-8. doi: 10.1016/j.amjcard.2004.09.036. PMID 15670547
- [Background] Sarrafzadegan N, Talaei M, Sadeghi M, Kelishadi R, Oveisgharan S, Mohammadifard N, Sajjadieh AR, Kabiri P, Marshall T, Thomas GN, Tavasoli A. The Isfahan cohort study: rationale, methods and main findings. J Hum Hypertens. 2011 Sep;25(9):545-53. doi: 10.1038/jhh.2010.99. Epub 2010 Nov 25. PMID 21107436
- [Background] Sanson-Fisher RW, Bonevski B, Green LW, D'Este C. Limitations of the randomized controlled trial in evaluating population-based health interventions. Am J Prev Med. 2007 Aug;33(2):155-61. doi: 10.1016/j.amepre.2007.04.007. PMID 17673104
- [Background] Relton C, Torgerson D, O'Cathain A, Nicholl J. Rethinking pragmatic randomised controlled trials: introducing the "cohort multiple randomised controlled trial" design. BMJ. 2010 Mar 19;340:c1066. doi: 10.1136/bmj.c1066. No abstract available. PMID 20304934
- [Derived] Dagenais GR, Pais P, Gao P, Roshandel G, Malekzadeh R, Joseph P, Yusuf S. Fixed dose combination therapies in primary cardiovascular disease prevention in different groups: an individual participant meta-analysis. Heart. 2023 Aug 24;109(18):1372-1379. doi: 10.1136/heartjnl-2022-322278. PMID 37258095
- [Derived] Roshandel G, Khoshnia M, Poustchi H, Hemming K, Kamangar F, Gharavi A, Ostovaneh MR, Nateghi A, Majed M, Navabakhsh B, Merat S, Pourshams A, Nalini M, Malekzadeh F, Sadeghi M, Mohammadifard N, Sarrafzadegan N, Naemi-Tabiei M, Fazel A, Brennan P, Etemadi A, Boffetta P, Thomas N, Marshall T, Cheng KK, Malekzadeh R. Effectiveness of polypill for primary and secondary prevention of cardiovascular diseases (PolyIran): a pragmatic, cluster-randomised trial. Lancet. 2019 Aug 24;394(10199):672-683. doi: 10.1016/S0140-6736(19)31791-X. PMID 31448738